CLINICAL TRIAL: NCT03170882
Title: A Phase 2, Randomized, Open-Label Study Comparing Oral Ixazomib/Dexamethasone and Oral Pomalidomide/Dexamethasone in Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study of Ixazomib, Given With Dexamethasone in Adults With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C16029; 2016-004742-28 (EudraCT Number); U1111-1188-2677 (Other: WHO); 2017/1235 (Registry Identifier: Norwegian Medicines Agency); N-20170083 (Registry Identifier: Danish Medicines Agency); 17/NW/0546 (Registry Identifier: NRES)
Record Dates: First submitted 2017-05-22; First posted 2017-05-31 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
Keywords: Drug therapy
MeSH Terms: interventions — ixazomib; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pomalidomide 4 mg + Dexamethasone 40 mg (Active Comparator): Pomalidomide 4 mg, capsules, orally, once daily on Days 1 to 21 of each 28-day cycle, plus dexamethasone 40 mg, (or 20 mg if participant is aged >=75 years), tablets, orally, once daily on Days 1, 8, 15, and 22 of each 28-day cycle until disease progression, unacceptable toxicity, withdrawal of consent, or sponsor termination of study up to 2 years.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone
- Ixazomib 4 mg + Dexamethasone 20 mg (Experimental): Ixazomib 4 mg as starting dose, capsules, orally, once daily on Days 1, 8, and 15 of each 28-day cycle, with escalation to 5.5 mg at the start of Cycle 2 for participants who tolerated the 4 mg dose in Cycle 1, plus dexamethasone 20 mg (or 10 mg if participant is aged >=75 years), tablets, orally, once daily on Days 1, 2, 8, 9, 15, 16, 22, and 23 of every 28-day cycle until disease progression, unacceptable toxicity, withdrawal of consent, or sponsor termination of study up to 2 years.
  Interventions: Drug: Ixazomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
  Other Names: NINLARO; MLN9708
  Arms: Ixazomib 4 mg + Dexamethasone 20 mg
Drug: Pomalidomide — Pomalidomide capsules
  Arms: Pomalidomide 4 mg + Dexamethasone 40 mg
Drug: Dexamethasone — Dexamethasone tablets

SUMMARY:
The main aim of this study is to learn if ixazomib, given with dexamethasone, stops the cancer from getting worse in people with relapsed or refractory multiple myeloma. It will be compared to another medicine called pomalidomide, given with dexamethasone with people with the same condition. Relapsed means the previous cancer treatment stopped working, over time. Refractory means they did not respond to previous cancer treatment. Another aim is to check for side effects from the study medicines.

At the first visit, the study doctor will check who can take part. Participants who can take part will be picked for 1 of 2 treatments by chance.

* Ixazomib capsules, given with dexamethasone tablets
* Pomalidomide capsules, given with dexamethasone tablets

All participants will take their study medicine on specific days during a 28-day cycle.

The 1st dose of study medicines in each 28-day cycle will take place in the clinic, The other doses of the study medicines will be taken at home. This will happen for 6 cycles. After this, all study medicines will be taken at home.

After treatment, participants will visit the clinic every 12 weeks for a check-up.

If participants cannot attend their clinic for an important reason (for example, due to the COVID-19 pandemic), the clinic will make alternative arrangements using their local procedures.

DETAILED DESCRIPTION:
The drug being tested in this study is called Ixazomib. Ixazomib is being tested to treat people who have relapsed and/or refractory multiple myeloma (RRMM). This study will compare the efficacy and safety in participants who take ixazomib and dexamethasone to pomalidomide and dexamethasone. It is an open-label, Phase 2 study.

The study will enroll approximately 120 participants. Participants will receive:

* Ixazomib 4 mg + dexamethasone 20 mg (or 10 mg if participant is aged >=75 years) OR
* Pomalidomide 4 mg + dexamethasone 40 mg (or 20 mg if participant is aged >=75 years)

All participants will be asked to take either ixazomib plus dexamethasone (in cases where only 4 mg tablets for dexamethasone are available, the following dexamethasone schedule is recommended for participants aged >=75 years: 12 mg dexamethasone will be given on Days 1, 8, 15, and 22 of every 28-day cycle; and 8 mg dexamethasone will be given on Days 2, 9, 16, and 23 of every 28-day cycle) or pomalidomide 4 mg + dexamethasone 40 mg at recommended doses.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is approximately 28 months after the first participant enters the study.

Participants will make multiple visits to the clinic, and will be contacted for progression free-survival (PFS) follow-up, in case of study drug discontinuation for up to 4 years from first dose administration. After disease progression, participants will be followed-up for overall survival (OS) every 12 weeks until death or up to 4 years.

Alternative methods for administering study procedures/assessments may be considered when it is not possible for the participants to come to the study site due to extenuating circumstances (e.g., due to the COVID-19 pandemic).

ELIGIBILITY:
Inclusion Criteria:

1. Must have a confirmed diagnosis of multiple myeloma (MM) requiring therapy according to International Myeloma Working Group (IMWG) criteria.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
3. Must have had a relapse or progressive disease (PD) after having received 2 or more prior lines of systemic therapy. Note: A line of therapy is defined as 1 or more cycles of a planned treatment program; this may consist of 1 or more planned cycles of single-agent therapy or combination therapy, as well as a sequence of treatments administered in a planned manner. For example, a planned treatment approach of induction therapy followed by autologous stem cell transplantation (SCT), followed by maintenance is considered 1 line of therapy. Typically each line of therapy is separated by PD. Discussion with the medical monitor may help clarify the number of lines of therapy that a prospective study participant had.
4. Must be refractory to lenalidomide, defined as having received at least 2 consecutive cycles of lenalidomide as a single agent or within a lenalidomide-containing regimen and having had PD during treatment with or within 60 days after the last dose of lenalidomide. The starting dose of lenalidomide should have been 25 mg (or as low as 10 mg in the case of renal function impairment or other safety concern), and the final dose should have been a minimum of 10 mg.
5. Must have received at least 2 consecutive cycles of a bortezomib- or carfilzomib-containing regimen, and either:

   * Achieved at least a partial response (PR) and did not have PD during treatment with or within 60 days after the last dose of bortezomib or carfilzomib, OR
   * Had bortezomib and/or carfilzomib intolerance (defined as discontinuation because of drug-related adverse events [AEs] before completion of the planned treatment course) without PD before the start of the next regimen.
6. Must have measurable disease defined by:

   * Serum M-protein >=1 g/dL (>=10 g/L), OR
   * Urine M-protein >=200 mg/24 hours and must have documented MM isotype by immunofixation (central laboratory).
7. Suitable venous access for the study-required blood sampling, including pharmacokinetic (PK) sampling.
8. Recovered (that is, less than or equal to [<=] Grade 1 nonhematologic toxicity) from the reversible effects of prior anticancer therapy.
9. Must be willing and able to adhere to pomalidomide-related risk mitigation activities if randomized to the pom+dex arm (example, Risk Evaluation and Mitigation Strategies [REMS], pregnancy prevention programs).

Exclusion Criteria:

1. Prior allogenic bone marrow transplantation in any prior line of therapy or prior autologous SCT in the last prior line of therapy- unless the autologous SCT was performed a year or more before disease progression.
2. Diagnosed with or treated for another malignancy within 2 years before randomization, or previously diagnosed with another malignancy and have any evidence of residual, persistent, or recurrent disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
3. Diagnosis of smoldering MM, Waldenström's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome, plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome.
4. Peripheral neuropathy Grade 1 with pain or Grade 2 or higher peripheral neuropathy of any cause on clinical examination during the Screening period.
5. Treatment with any investigational products or with chimeric or fully human monoclonal antibodies within 30 days before randomization, systemic anticancer therapy or radiotherapy within 14 days before randomization (Note: "spot" radiation for areas of pain is permitted), and major surgery within 14 days before randomization.
6. Known gastrointestinal disease or gastrointestinal procedure that could interfere with the oral absorption or tolerance of study therapy, including difficulty swallowing.
7. Serious infection requiring parenteral antibiotic therapy or any other serious infection within 14 days before randomization.
8. Central nervous system involvement with MM (by clinical symptoms and signs).
9. Ongoing or active systemic infection, known human immunodeficiency virus-ribonucleic acid (RNA) positive, known hepatitis B surface antigen seropositive, or known hepatitis C virus-RNA positive.
10. Systemic treatment with strong cytochrome P-450 3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital) or use of St. John's wort within 14 days before randomization.
11. Admission or evidence of illicit drug use, drug abuse, or alcohol abuse.
12. History of severe cutaneous reactions, including hypersensitivity reactions such as Stevens-Johnson syndrome (SJS), Toxic Epidermal Necrolysis (TEN), and Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS), in the context of treatment with lenalidomide or thalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (111):
- United States (10):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Lynn Cancer Institute, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Michigan State University, Lansing, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - San Juan Oncology Associates, Farmington, New Mexico
  - University of Toledo Medical Center, Toledo, Ohio
- Australia (5):
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Royal Adelaide Hospital, Adelaide
- Belgium (2):
  - GasthuisZusters Antwerpen, Wilrijk, Antwerpen
  - AZ St Jan Brugge Oostende AV, Bruges
- Canada (2):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Lakeridge Health Center, Ottawa, Ontario
- Czechia (7):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Kralovehradeck Kraj
  - University Hospital Olomouc, Olomouc, Olomouck Kraj
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Praha, Hlavni Mesto
  - Vseobecna fakultni nemocnice v Praze, Prague, Praha, Hlavni Mesto
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Plzen, Plzen Lochotin
- Denmark (2):
  - Aalborg Universitetshospital, Aalborg, North Denmark
  - Regionshospitalet Holstebro, Holstebro
- France (18):
  - Centre Antoine Lacassagne Centre Regional de Lutte Contre Le Cancer, Nice, Alpes-Maritimes
  - CHRU Dijon Complexe Du Bocage, Dijon, Cote-d'Or
  - CHRU de Brest - Hopital Morvan, Brest, Finistere
  - CHRU Nancy, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre Hospitalier Bretagne Atlantique Vannes, Vannes, Morbihan
  - Centre Hospitalier Le Mans, Le Mans, Sarthe
  - Groupe Hospitalier du Havre, Montivilliers, Seine-Maritime
  - CHU Amiens Hopital Sud, Amiens
  - Centre Hospitalier Fleyriat, Bourg-en-Bresse
  - Centre Hospitalier (CH) William Morey, Chalon-sur-Saône
  - Hospital d Instructions des Armees Percy, Clamart
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Centre Jean Bernard Clinique Victor Hugo, Le Mans
  - Centre Hospitalier Regional d'Orleans, Orléans
  - Centre Hospitalier de Perigueux, Périgueux
  - CHRU de Poitiers La Miletrie, Poitiers
  - CHRU Rennes, Rennes
  - Centre Henri Becquerel, Rouen
- Germany (4):
  - Uberortliche Gemeinschaftspraxis Pasing und Furstenfeldbruck, München, Bavaria
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Asklepios Klinik Altona, Hamburg
  - Universitatsklinikum Tubingen, Tübingen
- Greece (6):
  - University General Hospital of Patras, Pátrai, Achaia
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Evangelismos General Hospital of Athens, Athens
  - Alexandra Hospital, Athens
  - University General Hospital of Ioannina, Ioannina
  - Theageneio Anticancer Oncology Hospital of Thessaloniki, Thessaloniki
- Israel (5):
  - Soroka University Medical Centre, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Corporation, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
- Italy (17):
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna, Emilia-Romagna
  - Ospedale Santa Maria Delle Croci, Ravenna, Emilia-Romagna
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Ospedale Infermi di Rimini, Rimini, Emilia-Romagna
  - Fondazione del Piemonte per lOncologia (IRCCS), Candiolo, Piedmont
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano, Piedmont
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Turin, Piedmont
  - Centro Di Riferimento Oncologico Della Basilicata, Rionero in Vulture, PZ
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro, The Marches
  - Centro Di Riferimento Oncologico, Aviano
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia, Brescia
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori IRST, Meldola
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Ospedale Santa Maria Della Misericordia, Udine
  - Azienda ULSS 6 Vicenza, Vicenza
- Netherlands (2):
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - Zuyderland Medisch Centrum, Sittard
- Norway (5):
  - Oslo Universitetssykehus HF Rikshospitalet, Oslo, Oppland
  - Haukeland Universitetssykehus, Bergen
  - Forde Sentralsjukehus, Førde
  - Stavanger Universitetssykehus, Stavanger
  - St Olavs Hospital, Trondheim
- Russia (5):
  - Kirov Research Institute of Haematology and Blood Transfusion, Kirov
  - Moscow Clinical Scientific Center, Moscow
  - City Clinical Hospital n a S P Botkin, Moscow
  - City Clinical Hospital # 40, Moscow
  - Samara State Medical University, Samara
- Spain (3):
  - Hospital Universitario Infanta Leonor, Madrid, Madrid, Communidad Delaware
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (3):
  - Helsingborg Lasarett, Helsingborg, Skåne County
  - Sodra Alvsborgs Sjukhus Boras, Borås
  - Norrlands Universitetssjukhus, Umeå
- Turkey (Türkiye) (6):
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Ankara
  - Gazi University Medical Faculty Gazi Hospital, Ankara
  - Ankara University Medical Faculty Cebeci Hospital, Ankara
  - Dokuz Eylul University Medical Faculty, Izmir
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Erciyes Universitesi Tip Fakultesi Hastanesi, Kayseri
- United Kingdom (9):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Betsi Cadwaladr University Health Board, Bodelwyddan, Denbighshire-SirDdinbych
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Kent and Canterbury Hospital, Canterbury, Kent
  - GenesisCare Oxford, Oxford, Oxfordshire
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - Leicester Royal Infirmary, Leicester
  - Singleton Hospital, Swansea
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Dimopoulos MA, Schjesvold F, Doronin V, Vinogradova O, Quach H, Leleu X, Montes YG, Ramasamy K, Pompa A, Levin MD, Lee C, Mellqvist UH, Fenk R, Demarquette H, Sati H, Vorog A, Labotka R, Du J, Darif M, Kumar S. Oral ixazomib-dexamethasone vs oral pomalidomide-dexamethasone for lenalidomide-refractory, proteasome inhibitor-exposed multiple myeloma: a randomized Phase 2 trial. Blood Cancer J. 2022 Jan 24;12(1):9. doi: 10.1038/s41408-021-00593-2. PMID 35075109
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/5f6b60204db2bf003ab49572

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 54 investigative sites in Australia, Turkey, Czech Republic, France, Germany, Italy, Netherlands, Norway, Spain, Israel, United Kingdom, Sweden, Greece, and Russian Federation from 01 August 2017 up to 26 November 2021.
Pre-assignment Details: Participants with a diagnosis of relapsed and/or refractory multiple myeloma (RRMM) who received at least 2 prior lines of therapy were enrolled in 2:3 ratio to receive pomalidomide + dexamethasone or ixazomib + dexamethasone in this study.
Period: Overall Study
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Started | 49 | 73
Treated: Safety Population (Safety Population included all participants who received at least 1 dose of any study drug.) | 47 | 72
ITT PRO Population (Intent-to-Treat Patient Reported Outcomes (ITT PRO) Population included participants with a measurement at study entry and at least one post study entry measurement for at least 1 subscale on all 3 questionnaires (EORTC QLQ-C30, EORTC QLQ-MY20 and EQ-5D-5L).) | 45 | 70
Completed | 0 | 0
Not Completed | 49 | 73
Not completed — Death | 17 | 29
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Reason not Specified | 28 | 36

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg | Total
Number analyzed (Participants) | 49 | 73 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (8.33) | 70.6 (8.60) | 69.4 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 38 | 61
  Male | 26 | 35 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 42 | 65 | 107
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 46 | 69 | 115
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 8 | 15 | 23
  Norway | 7 | 8 | 15
  Italy | 9 | 5 | 14
  France | 3 | 9 | 12
  Ireland | 3 | 6 | 9
  Germany | 1 | 6 | 7
  Turkey | 4 | 3 | 7
  Spain | 2 | 4 | 6
  Israel | 3 | 2 | 5
  Czechia | 1 | 3 | 4
  Netherlands | 2 | 2 | 4
  Greece | 0 | 3 | 3
  Sweden | 2 | 1 | 3
  Australia | 4 | 6 | 10
Baseline Height [Mean (Standard Deviation); unit: cm] | 166.59 (8.740) | 165.01 (10.475) | 165.65 (9.808)
Baseline Weight [Mean (Standard Deviation); unit: kg] | 75.75 (16.160) | 74.36 (17.426) | 74.92 (16.875)
Baseline Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.864 (0.2203) | 1.837 (0.2430) | 1.848 (0.2336)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS: Time from randomization to first occurrence of confirmed progressive disease (PD) as assessed by investigator by International Myeloma Working Group(IMWG) response criteria/death from any cause, whichever occurs first. PD requires following: Increase of >=25 % from nadir in: Serum M component (increase must be >=0.5 gram per deciliter [g/dl]); Urine M-component (increase must be >=200 milligram [mg]/24-hour); In participants without measurable serum and urine M-protein levels difference between involved and uninvolved free light chain (FLC) increase of >10 mg/dl; In participants without measurable serum and urine M protein levels and without measurable disease by FLC level: bone marrow plasma cell percentage must be >=10%; Development of new/increase in size of existing bone lesions/soft tissue plasmacytomas; development of hypercalcemia (>11.5mg/dL corrected serum calcium) attributed solely to plasma cell proliferative disease.
Time Frame: From date of randomization until first occurrence of confirmed disease progression or death due to any cause, whichever occurs first (Up to approximately 3 years)
Population: ITT Population included all participants who were randomized. Participants without documentation of PD were censored at the date of last response assessment that is stable disease (SD) or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 49 | 73
months | 4.8 [3.745 to 8.542] | 7.1 [3.943 to 11.138]
Statistical Analysis 1: Comparison: Pomalidomide 4 mg + Dexamethasone 40 mg vs Ixazomib 4 mg + Dexamethasone 20 mg; Test type: Superiority; p = 0.477, Log Rank; Hazard Ratio (HR) = 0.847, 95% CI 2-sided [0.535 to 1.341] — HR obtained by unadjusted Cox's proportional hazard regression model stratified by age,international staging system(ISS),prior lines of therapy. HR<1 was deemed to indicate better PFS in Ixazomib+Dexamethasone arm over Pomalidomide+Dexamethasone arm

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause, up to 3 years are reported.
Time Frame: From date of randomization to death due to any cause (Up to approximately 3 years)
Population: ITT Population included all participants who were randomized. Participants without documented death at the time of analysis were censored at the date last known to be alive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 49 | 73
months | NA [13.963 to NA] — Median and upper limit of 95% confidence interval (CI) were not estimable due to low number of participants with events. | 18.8 [10.973 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Pomalidomide 4 mg + Dexamethasone 40 mg vs Ixazomib 4 mg + Dexamethasone 20 mg; Test type: Superiority; p = 0.265, Log Rank; Hazard Ratio (HR) = 1.427, 95% CI 2-sided [0.761 to 2.677] — HR obtained by unadjusted Cox's proportional hazard regression model stratified by age, ISS and prior lines of therapy. HR <1 was deemed to indicate longer survival time in Ixazomib + Dexamethasone arm as compared to Pomalidomide + Dexamethasone arm

3. Secondary Outcome: Percentage of Participants With Overall Response
Description: Overall Response Rate (ORR) was defined as the percentage of participants who achieved partial response (PR), very good partial response (VGPR), or complete response (CR) based on laboratory results and IRC assessment using modified IMWG criteria. PR: >=50% reduction of serum M protein + reduction in 24-hour urinary M protein by >=90% or to <200 mg/24-hour; if M protein is not measurable, >=50% decrease in difference between involved and uninvolved FLC levels is required; if not measurable by FLC, >=50% reduction in bone marrow plasma cells, when baseline value >=30% and; if present at baseline, >=50% reduction in size of soft tissue plasmacytomas is required. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein + urine M-protein level <100 mg/24-hour. CR: negative immunofixation on serum + urine; disappearance of soft tissue plasmacytomas; <5 % plasma cells in bone marrow.
Time Frame: From date of randomization until first documentation of CR, VGPR or PR (Up to approximately 3 years)
Population: ITT Population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 49 | 73
percentage of participants | 41 [27 to 56] | 38 [27 to 50]
Statistical Analysis 1: Comparison: Pomalidomide 4 mg + Dexamethasone 40 mg vs Ixazomib 4 mg + Dexamethasone 20 mg; Test type: Superiority; p = 0.634, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.43 to 1.90] — OR was based on logistic regression model with treatment group as categorical predictor variable and age, ISS and prior lines of therapy. OR >1 was deemed to indicate better response in Ixazomib+Dexamethasone arm over Pomalidomide+Dexamethasone arm

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR: Time from first documentation of CR/PR/VGPR to first documentation of PD. Per IMWG criteria, PR:>=50% reduction of serum M protein+reduction in 24-hour urinary M protein by >=90% to <200 mg/24-hour or >=50% decrease in difference between involved and uninvolved FLC levels/ >=50% reduction in bone marrow plasma cells, if >=30% at Baseline/ >=50% reduction in size of soft tissue plasmacytomas. VGPR: serum+urine M-protein detectable by immunofixation but not on electrophoresis/ >=90% reduction in serum M-protein + urine M-protein level <100 mg/24-hour. CR:negative immunofixation on serum + urine+disappearance of soft tissue plasmacytomas+<5% plasma cells in bone marrow. PD:serum M-component increase >=0.5 g/dl or urine M-component increase >=200 mg/24-hour/ difference between involved and uninvolved FLC levels increase >10 mg/dl or bone marrow plasma cell >=10%/development of new/ increase in size of existing bone lesions or soft tissue plasmacytoma or development of hypercalcemia.
Time Frame: From date of first documentation of CR, VGPR or PR until first occurrence of confirmed disease progression or death due to any cause, whichever occurs first (Up to approximately 3 years)
Population: Response Evaluable Population included all participants with multiple myeloma who had documentation of a confirmed PR, or PR/VGPR/CR. Only responders were reported for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 20 | 28
months | 14.3 [3.713 to NA] — Upper limit of 95% CI was not estimable due to low number of responders with events. | 14.8 [10.152 to 19.614]

5. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from randomization to the first documentation of PR/VGPR/CR. Per IMWG criteria, PR: >=50% reduction of serum M protein + reduction in 24-hour urinary M protein by >=90% or to <200 mg/24-hour; if M-protein is not measurable, >=50% decrease in difference between involved and uninvolved FLC levels is required; if not measurable by FLC, >=50% reduction in bone marrow plasma cells, when Baseline value >=30% and; if present at Baseline, >=50% reduction in size of soft tissue plasmacytomas is required. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein + urine M-protein level <100 mg/24-hour. CR: negative immunofixation on serum + urine; disappearance of soft tissue plasmacytomas; <5% plasma cells in bone marrow.
Time Frame: From date of randomization until first documentation of CR, VGPR or PR (Up to approximately 3 years)
Population: Response Evaluable Population included all participants with multiple myeloma who had documentation of a confirmed PR, or PR/VGPR/CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 49 | 73
months | 1.1 [0.953 to 2.037] | 2.0 [1.906 to 2.858]
Statistical Analysis 1: Comparison: Pomalidomide 4 mg + Dexamethasone 40 mg vs Ixazomib 4 mg + Dexamethasone 20 mg; Test type: Superiority; Hazard Ratio (HR) = 0.556, 95% CI 2-sided [0.288 to 1.073] — HR was obtained by unadjusted Cox's proportional hazard regression model stratified by age, ISS, prior lines of therapy. HR >1 was deemed to indicate quicker response time in Ixazomib + Dexamethasone arm over Pomalidomide + Dexamethasone arm

6. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from the date of randomization to first documentation of PD. Per IMWG criteria, PD required 1 of the following: Increase of >=25% from nadir in: Serum M-component (increase must be >=0.5 g/dl; Urine M-component (increase must be >=200 mg/24-hour); In participants without measurable serum and urine M-protein levels difference between involved and uninvolved FLC levels increase of >10 mg/dl; In participants without measurable serum and urine M protein levels and without measurable disease by FLC level: Bone marrow plasma cell percentage must be >=10%; Development of new or increase in size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (>11.5 mg/dL corrected serum calcium) attributed solely to plasma cell proliferative disease.
Time Frame: as for outcome 1
Population: ITT Population included all participants who were randomized. Participants without documentation of PD at the time of analysis are censored at the date of last response assessment that is SD or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 49 | 73
months | 5.1 [3.844 to 12.485] | 8.4 [5.684 to 13.306]
Statistical Analysis 1: Comparison: Pomalidomide 4 mg + Dexamethasone 40 mg vs Ixazomib 4 mg + Dexamethasone 20 mg; Test type: Superiority; p = 0.459, Log Rank; Hazard Ratio (HR) = 0.830, 95% CI 2-sided [0.506 to 1.361] — HR: obtained by unadjusted Cox's proportional hazard regression model stratified by age,ISS,prior lines of therapy. HR<1 was deemed to indicate better disease progression prevention in Ixazomib+Dexamethasone arm over Pomalidomide+Dexamethasone arm

7. Secondary Outcome: Health-Related Quality of Life (HRQOL) Based on European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire- Core 30 (EORTC QLQ-C30) Physical Domain Score
Description: The EORTC QLQ-C30 contains 30 items across 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status/quality of life (QOL) scale. The physical domain consisted of 5 items covering participant's daily physical activities on a scale from 1 (not at all) to 4 (very much). Raw scores were linearly transformed to a total score between 0-100, with a high score indicating better physical functioning.
Time Frame: Baseline and End of Treatment (Up to 28 cycles, each cycle was of 28 days)
Population: ITT PRO Population included participants with a measurement at study entry and at least one post study entry measurement for at least 1 subscale on all 3 questionnaires (EORTC QLQ-C30, EORTC Multiple Myeloma Module 20 [QLQ-MY20] and EuroQol 5-Dimensional Health Questionnaire [EQ-5D-5L]). Number analyzed are the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 45 | 70
score on a scale
  Baseline | 67.0 (21.97) | 67.9 (22.08)
  End of Treatment: number analyzed (Participants) | 28 | 42
  End of Treatment | 52.4 (28.03) | 56.5 (26.10)

8. Secondary Outcome: HRQOL Based on EORTC QLQ-C30 SubScale Score
Description: The EORTC QLQ-C30 contains 30 items across 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial difficulties) and a QOL scale. Most of the 30 items had 4 response levels (not at all, a little, quite a bit, and very much), with 2 questions relying on a 7-point numeric rating scale. Each subscale raw score were linearly transformed to a total score between 0 to 100. For the functional scales and the global health status/QOL scale, higher scores represent better QOL; for the symptom scales, lower scores represent better QOL. The Physical domain of the functional subscale is reported in the secondary outcome measure 7.
Time Frame: Baseline and End of Treatment (Up to 28 cycles, each cycle was of 28 days)
Population: ITT PRO Population included participants with a measurement at study entry and at least one post study entry measurement for at least 1 subscale on all 3 questionnaires (EORTC QLQ-C30, EORTC QLQ-MY20 and EQ-5D-5L). Number analyzed are the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 45 | 70
score on a scale
  Global Health Status/QoL: Baseline | 57.0 (20.72) | 60.8 (21.16)
  Global Health Status/QoL: End of Treatment: number analyzed (Participants) | 27 | 42
  Global Health Status/QoL: End of Treatment | 47.8 (19.56) | 48.2 (19.61)
  Role (Functional Scale): Baseline | 67.4 (28.42) | 67.9 (29.67)
  Role (Functional Scale): End of Treatment: number analyzed (Participants) | 28 | 42
  Role (Functional Scale): End of Treatment | 47.6 (27.86) | 49.2 (27.04)
  Emotional (Functional Scale): Baseline | 74.9 (21.19) | 83.1 (21.70)
  Emotional (Functional Scale): End of Treatment: number analyzed (Participants) | 28 | 42
  Emotional (Functional Scale): End of Treatment | 67.6 (25.19) | 72.8 (22.62)
  Cognitive(Functional Scale): Baseline | 79.6 (20.38) | 84.0 (20.74)
  Cognitive (Functional Scale): End of Treatment: number analyzed (Participants) | 28 | 42
  Cognitive (Functional Scale): End of Treatment | 69.6 (27.61) | 77.4 (22.64)
  Social (Functional Scale): Baseline | 72.2 (29.94) | 75.7 (27.02)
  Social (Functional Scale): End of Treatment: number analyzed (Participants) | 28 | 42
  Social (Functional Scale): End of Treatment | 63.1 (27.35) | 69.8 (24.76)
  Fatigue (Symptom Scale): Baseline | 60.0 (22.89) | 61.0 (23.07)
  Fatigue (Symptom Scale): End of Treatment: number analyzed (Participants) | 28 | 42
  Fatigue (Symptom Scale): End of Treatment | 50.8 (25.02) | 50.3 (25.77)
  Nausea/Vomiting (Symptom Scale): Baseline | 96.7 (8.41) | 94.8 (11.54)
  Nausea/Vomiting (Symptom Scale): End of Treatment: number analyzed (Participants) | 28 | 42
  Nausea/Vomiting (Symptom Scale): End of Treatment | 88.7 (15.75) | 92.9 (16.52)
  Pain (Symptom Scale): Baseline | 61.1 (30.77) | 65.2 (24.70)
  Pain (Symptom Scale): End of Treatment: number analyzed (Participants) | 28 | 42
  Pain (Symptom Scale): End of Treatment | 51.2 (26.42) | 53.2 (28.33)
  Dyspnea (Symptom Scale): Baseline | 25.2 (28.56) | 19.0 (25.74)
  Dyspnea (Symptom Scale): End of Treatment: number analyzed (Participants) | 28 | 42
  Dyspnea (Symptom Scale): End of Treatment | 40.5 (30.57) | 24.6 (26.61)
  Insomnia (Symptom Scale): Baseline | 32.6 (29.72) | 29.5 (31.87)
  Insomnia (Symptom Scale): End of Treatment: number analyzed (Participants) | 28 | 42
  Insomnia (Symptom Scale): End of Treatment | 36.9 (34.35) | 29.4 (34.69)
  Appetite Loss (Symptom Scale): Baseline | 22.2 (27.52) | 14.3 (22.39)
  Appetite Loss (Symptom Scale): End of Treatment: number analyzed (Participants) | 28 | 42
  Appetite Loss (Symptom Scale): End of Treatment | 34.5 (34.52) | 23.0 (28.02)
  Constipation (Symptom Scale): Baseline | 13.3 (23.99) | 11.4 (20.37)
  Constipation (Symptom Scale): End of Treatment: number analyzed (Participants) | 28 | 42
  Constipation (Symptom Scale): End of Treatment | 25.0 (34.69) | 19.8 (29.50)
  Diarrhea (Symptom Scale): Baseline | 17.8 (23.14) | 16.7 (23.23)
  Diarrhea (Symptom Scale): End of Treatment: number analyzed (Participants) | 28 | 41
  Diarrhea (Symptom Scale): End of Treatment | 19.0 (26.34) | 16.3 (25.95)
  Financial Difficulties (Symptom Scale): Baseline | 22.2 (27.52) | 17.1 (25.85)
  Financial Difficulties (Symptom Scale): End of Treatment: number analyzed (Participants) | 28 | 42
  Financial Difficulties (Symptom Scale): End of Treatment | 16.7 (21.28) | 12.7 (22.03)

9. Secondary Outcome: HRQOL Based on EORTC Multiple Myeloma Module 20 (EORTC QLQ-MY20) Score
Description: The EORTC QLQ-MY20 has 20 items across 4 independent subscales, 2 symptoms scales (disease symptoms, side effects of treatment), and 2 functional subscales (body image, future perspective). Scores were averaged and transformed to 0-100 scale. Higher scores for the future perspective scale indicate better perspective of the future, for the body image scale indicate better body image and for the disease symptoms scale indicate higher level of symptomatology.
Time Frame: Baseline and End of Treatment (Up to 28 cycles, each cycle was of 28 days)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 45 | 70
score on a scale
  Disease Symptoms: Baseline | 73.2 (17.06) | 72.4 (21.31)
  Disease Symptoms: End of Treatment: number analyzed (Participants) | 28 | 41
  Disease Symptoms: End of Treatment | 73.5 (17.75) | 68.9 (23.09)
  Side Effects of Treatment: Baseline | 81.0 (13.45) | 81.4 (13.30)
  Side Effects of Treatment: End of Treatment: number analyzed (Participants) | 28 | 41
  Side Effects of Treatment: End of Treatment | 74.4 (17.84) | 77.8 (14.47)
  Body Image: Baseline | 81.5 (23.09) | 82.9 (23.90)
  Body Image: End of Treatment: number analyzed (Participants) | 28 | 41
  Body Image: End of Treatment | 75.0 (30.93) | 83.7 (23.71)
  Future Perspective: Baseline | 58.8 (23.29) | 67.5 (24.03)
  Future Perspective: End of Treatment: number analyzed (Participants) | 28 | 41
  Future Perspective: End of Treatment | 57.9 (28.26) | 64.0 (19.21)

10. Secondary Outcome: Number of Participants With Responses to HRQOL Based on 5-level Classification System of the EuroQol 5-Dimensional Health Questionnaire (EQ-5D-5L) Score
Description: EQ-5D-5L comprises of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, 5= extremely severe problems. Higher scores indicated greater levels of problems across the five dimensions.
Time Frame: End of Treatment (Up to 28 cycles, each cycle was of 28 days)
Population: ITT PRO Population included participants with a measurement at study entry and at least one post study entry measurement for at least 1 subscale on all 3 questionnaires (EORTC QLQ-C30, EORTC QLQ-MY20 and EQ-5D-5L). Overall number of participants analyzed are the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 27 | 41
Participants
  Mobility: 1 = I Have no Problems in Walking About | 5 | 9
  Mobility: 2 = I Have Slight Problems in Walking About | 6 | 12
  Mobility: 3 = I Have Moderate Problems in Walking About | 8 | 11
  Mobility: 4 = I Have Severe Problems in Walking About | 8 | 8
  Mobility: 5 = I am Unable to Walk About | 0 | 1
  Self-Care: 1 = I Have no Problems Washing or Dressing Myself | 13 | 21
  Self-Care: 2 = I Have Slight Problems Washing or Dressing Myself | 6 | 10
  Self-Care: 3 = I Have Moderate Problems Washing or Dressing Myself | 5 | 4
  Self-Care: 4 = I Have Severe Problems Washing or Dressing Myself | 3 | 4
  Self-Care: 5 = I am Unable to Wash or Dress Myself | 0 | 2
  Usual Activities: 1 = I Have no Problems Doing my Usual Activities | 4 | 10
  Usual Activities: 2 = I Have Slight Problems Doing my Usual Activities | 7 | 9
  Usual Activities: 3 = I Have Moderate Problems Doing my Usual Activities | 8 | 12
  Usual Activities: 4 = I Have Severe Problems Doing my Usual Activities | 7 | 7
  Usual Activities: 5 = I am Unable to do my Usual Activities | 1 | 3
  Pain/Discomfort: 1 = I Have no Pain or Discomfort | 3 | 8
  Pain/Discomfort: 2 = I Have Slight Pain or Discomfort | 5 | 10
  Pain/Discomfort: 3 = I Have Moderate Pain or Discomfort | 13 | 15
  Pain/Discomfort: 4 = I Have Severe Pain or Discomfort | 6 | 6
  Pain/Discomfort: 5 = I Have Extreme Pain or Discomfort | 0 | 2
  Anxiety/Depression: 1 = I Have no Pain or Discomfort | 6 | 19
  Anxiety/Depression: 2 = I Have no Pain or Discomfort | 8 | 13
  Anxiety/Depression: 3 = I Have no Pain or Discomfort | 11 | 6
  Anxiety/Depression: 4 = I Have no Pain or Discomfort | 2 | 1
  Anxiety/Depression: 5 = I Have no Pain or Discomfort | 0 | 2

11. Secondary Outcome: HRQOL Based on EuroQol Visual Analogue Scale (EQ VAS) Score
Description: The EQ VAS records the respondent's self-rated health on a 20 centimeter (cm), vertical, visual analogue scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). The scores from all dimensions were combined into a single index score that was reported, where higher score was better quality of life.
Time Frame: Baseline and End of Treatment (Up to 28 cycles, each cycle was of 28 days)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 45 | 70
score on a scale
  Baseline | 59.2 (20.96) | 64.4 (18.21)
  End of Treatment: number analyzed (Participants) | 27 | 41
  End of Treatment | 46.9 (19.07) | 55.9 (19.60)

12. Secondary Outcome: Health Care Utilization (HU): Number of Participants With at Least One Medical Encounter
Description: Healthcare resources used during medical encounters included hospitalizations, emergency room stays, or outpatient visits. A hospitalization was defined as at least 1 overnight stay in an Intensive Care Unit and/or non-Intensive Care Unit (acute care unit, palliative care unit, and hospice).
Time Frame: Up to approximately 3 years
Population: ITT Population included all participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 49 | 73
Participants
  Hospitalizations | 16 | 23
  Emergency Room Stays | 9 | 11
  Outpatient Visits | 29 | 32

13. Secondary Outcome: HU: Duration of Medical Encounters
Description: Duration of healthcare resources used during medical encounters including hospitalizations, emergency room stays, or outpatient visits was reported in days. A hospitalization was defined as at least 1 overnight stay in an Intensive Care Unit and/or non-Intensive Care Unit (acute care unit, palliative care unit, and hospice).
Time Frame: Up to approximately 3 years
Population: ITT Population included all participants who were randomized.
Measure: Median (Full Range); unit: days
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
Number analyzed (Participants) | 49 | 73
days
  Hospitalizations | 2.0 [1.0 to 6.0] | 1.0 [1.0 to 10.0]
  Emergency Room Stays | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Outpatient Visits | 4.0 [1.0 to 57.0] | 3.0 [1.0 to 34.0]

ADVERSE EVENTS:
Time Frame: From signing of the informed consent up to 30 days after last dose of the study drug (Up to approximately 4 years 3 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. All cause-mortality was collected for all randomized participants. Serious and other (non-serious) adverse events were collected for participants from Safety Population who received at least 1 dose of any study drug.
Arm/Group | Pomalidomide 4 mg + Dexamethasone 40 mg | Ixazomib 4 mg + Dexamethasone 20 mg
All-Cause Mortality (participants affected / at risk) | 17/49 | 29/73
Serious Adverse Events (participants affected / at risk) | 26/47 | 40/72
Other Adverse Events (participants affected / at risk) | 45/47 | 62/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide 4 mg + Dexamethasone 40 mg (N=47) | Ixazomib 4 mg + Dexamethasone 20 mg (N=72)
Pneumonia (Infections and infestations) | 10 | 9
Bronchitis (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
H1N1 influenza (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 2
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Enterobacter sepsis (Infections and infestations) | 1 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 2
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 3
Atrial tachycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Facial pain (General disorders) | 1 | 0
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Enterobacter test positive (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 0 | 1
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0
Sialodenitis (Infections and infestations) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide 4 mg + Dexamethasone 40 mg (N=47) | Ixazomib 4 mg + Dexamethasone 20 mg (N=72)
Diarrhoea (Gastrointestinal disorders) | 13 | 28
Nausea (Gastrointestinal disorders) | 7 | 12
Constipation (Gastrointestinal disorders) | 8 | 9
Vomiting (Gastrointestinal disorders) | 4 | 10
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 18 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 16
Neutropenia (Blood and lymphatic system disorders) | 20 | 1
Fatigue (General disorders) | 11 | 17
Asthenia (General disorders) | 8 | 4
Oedema peripheral (General disorders) | 2 | 10
Pyrexia (General disorders) | 7 | 4
Influenza like illness (General disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 7 | 7
Bronchitis (Infections and infestations) | 6 | 7
Urinary tract infection (Infections and infestations) | 6 | 4
Pneumonia (Infections and infestations) | 4 | 4
Nasopharyngitis (Infections and infestations) | 3 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 19
Dizziness (Nervous system disorders) | 4 | 5
Headache (Nervous system disorders) | 0 | 4
Tremor (Nervous system disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 5
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1
Insomnia (Psychiatric disorders) | 5 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Platelet count decreased (Investigations) | 4 | 9
Neutrophil count decreased (Investigations) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 5
Hypertension (Vascular disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT03170882/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03170882/SAP_001.pdf